CLINICAL TRIAL: NCT07230808
Title: A Pilot Feasibility Study of Digitally Delivered Modules Focused on Preventing the Development of Obesity During the First Year of Life Within an Existing Statewide Home Visitation Program
Brief Title: Digitally Delivered Child Obesity Prevention for Parents in Home Visiting Programs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB202501112; R34HL163373 (NIH)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Childhood Obesity Prevention
Keywords: childhood obesity; home visiting; parents; infants; nutrition education; eHealth; digital intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital intervention (Experimental): digitally delivered childhood obesity prevention intervention for parents
  Interventions: Behavioral: digital intervention + home visiting curriculum
- standard home visiting curriculum (Active Comparator): standard home visiting program for parents
  Interventions: Behavioral: Home visiting curriculum

INTERVENTIONS:
Behavioral: digital intervention + home visiting curriculum — Digitally delivered childhood obesity prevention intervention for parents called THRIVES (Teaching Healthy Routines in Very Early Stages) will be provided to complement the standard home visiting curriculum. Parents will complete digital content containing videos, text and checkpoint questions with goal setting during the first year of their child's life over a 12 month period. Assessments will be collected at baseline, 4, 6 and 12 months.
  Arms: Digital intervention
Behavioral: Home visiting curriculum — Parents will receive a standard home visiting curriculum delivered in person for at least 1 year during the project timeframe and complete assessments at baseline, 4, 6 and 12 months.
  Arms: standard home visiting curriculum

SUMMARY:
The goal of this clinical trial is to determine feasibility and acceptability of a digitally-based obesity prevention intervention for mothers of infants participating in a home visitation program.

The main questions it aims to answer are:

* What impact does the digitally based obesity prevention intervention for parents have on children's weight?
* What impact does the digitally based obesity prevention intervention have on mothers' feeding practices, child sleep, and child screen time? Researchers will compare the digital intervention to home visiting standard curriculum to see if the intervention results in larger improvements.

Participants will view several digital modules including videos on feeding, activity and family topics over the course of 1 year. They will complete questionnaires at the beginning of the study and again at 4, 6 and 12 months and their child will be weighed and measured at each time point.

DETAILED DESCRIPTION:
The first 1,000 days (conception to age 2) have been deemed a critical period for obesity prevention yet, effective, sustainable efforts are lacking. Current home visitation programs (HVP) targeting at-risk families for other child development related issues are a potential innovative opportunity for early childhood obesity prevention. The overall goal of the project is to reduce the prevalence of overweight and obesity in children under the age of 1 year thereby reducing obesity rates of older children and adults in the long term. Prior pilot work by members of the research team demonstrated feasibility of embedding an early childhood obesity prevention (ECHO) program in an existing home visitation program (HVP+) during an infant's first year of life.

Five obesity-associated behaviors (i.e., breastfeeding, introduction to solids, limiting juice, sleep routines, screen time) were emphasized through brief interactive lessons utilizing behavior change strategies and an ecological approach by providing linkages to community resources that support healthy behaviors. The pilot program was well received by families, mothers breastfed longer, infants had fewer nocturnal awakenings, were less likely to receive juice, and had a lower weight-for-length (WFL) z-score at 12 months. However, there is a critical need for alternative and innovative, consistent, and sustainable digital delivery methods especially during times when face-to-face home visits are not feasible. Qualitative interviews were conducted with home visitors (n=27) from Florida's (FL) Maternal, Infant Early Childhood Home Visitation (MIECHV) Program and revealed that they were highly receptive to using digital learning with at-risk families.

The specific aims of the proposed research are to a) Develop, refine, and conduct usability testing of early childhood obesity prevention digital learning modules with mothers participating in FL MIECHV; and b) Conduct a pilot RCT of a 12 month digitally-enhanced early childhood obesity prevention intervention (HVP+E), with 50 mother-infant pairs (25 HVP+E/25 standard HVP) participating in FL MIECHV to determine feasibility and acceptability of the HVP+E intervention and study recruitment, implementation and evaluation protocols; and obtain data on preliminary efficacy of the intervention on children's WFL z-scores (primary outcome), maternal feeding practices, child sleep and screen time (secondary outcomes).

Mother-infant dyads (n=50) enrolled in the Maternal, Infant Early Childhood Home Visitation (MIECHV) Program parentally or within one month of giving birth will be randomized to receive either the standard home visitation program (HVP) or the digitally delivered obesity prevention-enhanced home visitation program (HVP+E) for 1 year. HVP+E content will also be expanded to support mothers in engaging fathers and other family members in target behaviors. Mother-infant dyads will be assessed at study entry and at 4, 6 and 12 months. If efficacious, the intervention has potential for public health impact through early childhood obesity prevention in an underserved population, and dissemination through home visitation programs nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in or eligible for home visiting program
* Ages 16 years or older
* Speaks and reads English
* Has no chronic health condition affecting growth or development
* Has a singleton birth > 37 weeks gestation.

Exclusion Criteria:

* Child has a major malformation
* Child admitted to the NICU
* Child considered small for gestation age (SGA) and/or have a low birth weight (<2500 gms)
* Mother has a significant maternal morbidity (e.g. cancer) or hospitalization for psychiatric disorder in past 6 months
* Extended hospital stay for mom or infant > 5 days
* Unable to speak and read English.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Child Weight for Length | 0, 4, 6, 12 months
  Weight for Length (WFL) z-score. A z-score of 0 indicates a child is a the median for WFL. Scores above 0 indicate that a child has a higher WFL and may be at risk for overweight or obesity. Scores below 0 indicate that a child has a lower WFL and may be at risk for undernutrition.

SECONDARY OUTCOMES:
Structure and Control in Parent Feeding Questionnaire (SCFQ) | 0, 4, 6, 12 months
  The SCFQ contains questions related to structure and controlling parental feeding practices. The validated questionnaire has two subscales: 1) Structure (meal routines, feeding environment, etc.) and 2) Control (pressure to eat, restriction, etc.). Responses are captured on a 5-point Likert scale with 1 indicating "never" and 5 indicating "always." Higher scores indicate greater structure or control while lower scores indicate lower structure or control.
Baby's Basic Needs Questionnaire (BBNQ) | 0, 4, 6, and 12 months
  Feeding to soothe practices will be captured using the BBNQ which assesses infant's feeding history and extent to which mothers use feeding to soothe their infants. Responses are captured on a 5-point Likert scale (1=Never; 5=Always). Higher scores indicate more frequent use of feeding to soothe while lower scores indicate less use of feeding to soothe.
Feeding behaviors of parents (breastfeeding, timing of juice and solid food introduction) | 0, 4, 6 and 12 months
  Questions were adapted from the Beverage Intake Questionnaire, Preschool Version (BEVQ-PS), an instrument designed to assess the frequency of preschool children's intake of beverages, including 100% fruit juice. In the BEVQ-PS, parents report how often their child consumes specific beverages using responses options ranging from "Never" to "3 or more times per day." Higher responses indicate more frequent intake and lower responses indicate less frequent intake.
  Other measures were adapted from the National Survey of Children's Health (NSCH) questionnaire, which includes standardized items assessing infant feeding practices. Parents report the age at which their child was first given food other than breastmilk or formula or juice, using response options as follows: <1 month, 2-3 months, 4-5 months, 6-8 months, 9-11 months, or 12 months or older. Responses will be compared to current solid food and juice guidance.
Parental obesity prevention knowledge, attitudes, and behaviors | From date of randomization until date of completion of the digital modules, assessed up to 1 year.
  Checkpoint questions associated with digital intervention module topics will administered after parents complete the digital modules. These items evaluate parents' knowledge, attitudes, and intentions related to obesity-prevention behaviors, including feeding, sleep, screen time, and soothing practices. The questions are not part of a validated scale; responses are summarized descriptively based on accuracy of answers and qualitatively.
Dietary Screener Questionnaire | 0, 4, 6 and 12 months
  The 26-item Dietary Screener Questionnaire (DSQ) will be used to assess the frequency of consumption in the past month of selected foods and drinks. The DSQ captures intakes of fruits and vegetables, dairy/calcium, added sugars, whole grains/fiber, red meat, and processed meat. The DSQ can be interviewer-administered on paper or the web. Each of the 26 items on the screener was selected because of its relationship to one or more dietary factors of interest in dietary guidance.The scoring algorithms convert screener responses to estimates of dietary intake for fruits and vegetables (cup equivalents), dairy (cup equivalents), added sugars (tsp), whole grains (ounce equivalents), fiber (g), and calcium (mg). Responses to the red meat and processed meat questions may be used as qualitative indicators of intake frequency.
Activity and Screen time | 0, 4, 6 and 12 months
  Parent and Child activity and screen time questions are adapted from a combination of project developed items and from the Infant Feeding Practices Study II (IFPS-II) and the National Survey of Children's Health (NSCH). The questionnaires are not operationalized on a validated scale; responses are summarized descriptively.
Brief Infant Sleep Questionnaire | 0, 4, 6 and 12 months
  Infant sleep duration and awakenings are measured using the Brief Infant Sleep Questionnaire (BISQ). The BISQ does not equate to an overall score with minimum or maximum values. Individual sleep parameters are reported descriptively
Postnatal Edinburgh Depression Scale | 0, 4, 6 and 12 months
  The Edinburgh Postnatal Depression Scale (EPDS), a 10-item validated tool measuring symptoms of postpartum depression, will be used to screen/assess depression of parent. Each item is scored from 0 to 3, producing a total score ranging from 0 to 30. Higher scores indicate more severe depressive symptoms and lower scores indicate less depressive symptoms.
Family Social Support Questionnaire | 0, 4, 6 and 12 months
  The Multidimensional Scale of Perceived Social Support (MSPSS), a 12-item validated measure, will be used to assess social support of the parent and is scored from 1 to 7. Subscale and total mean scores also range from 1 to 7, with higher scores indicating greater perceived social support and lower scores indicating less perceived social support. Results are summarized using mean scores.
Perceived Stress Scale | 0, 4, 6 and 12 months
  The Perceived Stress Scale (PSS), a validated 10-item measure of perceived stress over the past month, will be used to assess stress of the parent. Each item is scored from 0 to 4, with a total score ranging from 0 to 40. Higher scores indicate greater perceived stress, and lower scores indicate lower perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Mobley, PhD, RD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No